CLINICAL TRIAL: NCT07041658
Title: Assessment of Nutritional Status of Critically Ill Children Admitted to Pediatric Intensive Care Units at Sohag University Hospitals
Brief Title: Nutritional Status of Critically Ill Children in Pediatric Intensive Care Units at Sohag University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Klara Boulis Anwar, Pediatric Specialist, Sohag University
Other Study IDs: Soh-Med-25-5--3MD
Record Dates: First submitted 2025-05-23; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Intensive Care Units

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate nutritional status of critically ill patients admitted to Pediatric Intensive Care Units (PICU) at Sohag University Hospital and its correlation with their outcome as regarding to need for mechanical ventilation, acquired infection, metabolic complications, and mortality.

DETAILED DESCRIPTION:
Nutrition is one of the important factors which affect morbidity and mortality in critically ill patients in pediatric intensive care units (PICU). Adequate and balanced nutrition is required not only to support physical growth and basic metabolic needs, but also to ensure proper organ function and sustain daily activities.

Nutritional status reflects the dynamic balance between nutrient availability, dietary intake, and the body's ability to absorb and utilize those nutrients in relation to an individual's specific needs.

Critical illness triggers significant metabolic and endocrine changes which are characterized by catabolism, insulin resistance, stress hyperglycemia and shifts in substrate utilization. These changes closely interact with disruptions in the autonomic and immune systems. Critically ill infants and children may have an increased metabolic need, which predisposes them to nutritional deterioration and malnutrition during illness.

The World Health Organization (WHO) defines malnutrition as " an acute or chronic nutritional status due to deficiency or excess energy, protein and micronutrient resulting in imbalance between nutrient intake and requirement that can negatively affect growth and development".

Malnutrition in critically ill patients is associated with decreased respiratory function, higher rate of nosocomial infections, secondary immunodeficiency, prolonged mechanical ventilation and prolonged hospitalization. It is also related to delayed wound healing process, impairment in gastrointestinal functions, thus increased morbidity and mortality.

The American and European Society of Parenteral and Enteral Nutrition guidelines recommend that nutritional status should be evaluated on admission to the PICU to identify children at risk and to provide nutrition support in the PICU.

Enteral feeding approach has been preferred to be started within the first 24-48 hours after admission to the PICU, if there are no contraindications for enteral nutrition. Early initiation of enteral feeding have been associated with improved clinical outcomes as regard morbidity and mortality. Metabolic demands must be determined by calculating energy consumption.

Malnutrition at PICU admission is frequent (15-25% prevalence rates) in developing countries. A study published in 2022 on the nutritional status of critically ill children in one Egyptian PICU found that malnutrition rate can be around 30%. However, the data on nutritional status in Egyptian PICUs is scarce especially in Upper Egypt. Therefore, assessment of nutritional status in our PICU can help in improving the outcome of critically ill children in terms of both morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All critically ill children who admitted in PICUs at Sohag University Hospital with age range from 1 month up to 16 years old.

Exclusion Criteria:

* Patient with recurrent admissions to the PICU during the specified study period, only the first admission will be included.
* Patient with PICU stay less than 48 hours.
* Patients referred with nutritional regimen or metabolic disease e.g. patients on ketogenic diet and patients with inborn errors of metabolism.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: critically ill children who admitted in PICUs at Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
need for mechanical ventilation | one week following PICU admission
acquired infection | one week following PICU admission
mortality | one week following PICU admission

IPD SHARING:
Plan to Share IPD: Undecided